CLINICAL TRIAL: NCT02677064
Title: Observational Study to Identify Barriers to Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Newly Diagnosed and Relapsed Acute Leukemia, Myelodysplastic Syndrome and Myelproliferative Neoplasms
Brief Title: Identify Barriers to Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Newly Diagnosed and Relapsed Acute Leukemia
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-024
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Acute Leukemia; Newly Diagnosed; Relapsed
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; Identify Barriers; 16-024
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Patients with Acute Leukemia (Arm A): Follow patients throughout their journey and identify prospectively the reasons why patients did not proceed to HCT when deemed appropriate and eligible.
  Interventions: Other: assessments
- Patients with MDS and MPN (Arm B): Follow patients throughout their journey and identify prospectively the reasons why patients did not proceed to HCT when deemed appropriate and eligible.
  Interventions: Other: assessments
- Patients with Acute Leukemia or MDS/MPN who Relapse After First Allografts (Arm C): Follow patients throughout their journey and identify prospectively the reasons why patients did not proceed to HCT when deemed appropriate and eligible.
  Interventions: Other: assessments

INTERVENTIONS:
Other: assessments — All laboratory assessments performed on this study represent standard of care at our institution. HLA allele typing is performed by the center's HLA laboratory according to standard typing procedures.

SUMMARY:
The investigators are doing this research study to assess the percentage of patients receiving stem cell transplantation for the type of blood cancer you have. They want to know how many patients get a transplant and why some patients do get a transplant while others do not. Also they want to explore why some patients elect not to undergo stem cell transplantation, when it is recommended by their physicians.

DETAILED DESCRIPTION:
Additional Arms have been added for MSK patients only. Patients with MDS and MPN Patients with Post-transplant Relapse of Acute Leukemia, MDS or MPN

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or relapsed acute leukemia. Patients undergoing reinduction due to primary induction failure are also eligible. Patients with acute leukemia will be enrolled to Arm A
* Patients with diagnosis of MDS, MPN and MDS/MPN overlap who meet any of the following criteria (based on NCCN guidelines):
* Clinically significant cytopenia of at least 2 cell lines affected; Hgb<10,
* Platelet<100,000, absolute neutrophil count<1000
* Bone marrow blasts >5% and any level of circulating blasts
* Evidence of disease progression or no response to hypomethylating agents/immunosuppressive treatment or a clinical trial.
* IPSS Intermediate-1 and higher
* IPSS-R intermediate and higher
* All cases of therapy related MDS with excess blasts
* In patients with Myelofibrosis: Low risk disease by DIPSS with either refractory, transfusion dependent anemia, circulating blasts cells greater than 2%; or adverse cytogenetics and any patient with DIPSS-intermidiate 1 and higher.
* Patients with acute leukemia or MDS/MPN who relapse after first allografts. Patients with post-transplant relapse will be enrolled to Arm C.
* Patients 18 years of age or older and 80 years of age or younger
* For the purposes of this protocol "relapse" is defined as re-emergence of the initial abnormal myeloid blast population (or blast equivalent) comprising 5% or more of marrow WBC or any amount prompting a therapeutic intervention targeting relapsed disease, including, but not limited to withdrawal of immunosuppression, targeted therapies, chemotherapy, etc.

Exclusion Criteria:

* Patients with polycythemia vera (PV) and essential thrombocytosis (ET)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute leukemia and MDS or MPN who are treated inpatient or outpatient by the Leukemia Service for induction or re-induction therapy (acute leukemia) or initiation of therapy (for MDS or MPN) will be seen by the Adult BMT Service.
Sampling Method: Non-Probability Sample
Enrollment: 1365 (Estimated)
Dates: Start 2016-02; Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
number of patients who proceed to transplant | 3 years
  determine whether an individual patient proceeded to HCT when he or she was considered eligible (based on NCCN guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Tamari, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/